CLINICAL TRIAL: NCT04640220
Title: The Effectiveness of Intra-articular Steroid Injection in Breast Cancer Survivors With Adhesive Capsulitis According to the Thickness of Axillary Capsulitis Thickness
Brief Title: Improvement of Range of Motion in Frozen Shoulder in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Dong Gyu Lee, Assistant professor, Yeungnam University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-07-064-002
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Breast Neoplasm; Shoulder Capsulitis; Range of Motion
MeSH Terms: conditions — Breast Neoplasms | interventions — Steroids

STUDY DESIGN:
Intervention Model Description: Adhesive capsulitis patients who underwent breast cancer operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adhesive capsulitis in breast cancer survivors (Experimental): Intra-articular steroid injection
  Interventions: Procedure: Intra-articular steroid injection

INTERVENTIONS:
Procedure: Intra-articular steroid injection — Ultrasound-guided Gleno-humeral joint steroid (Triamcinolone 40mg with 0.5% lidocaine ) injection

SUMMARY:
The prevalence of shoulder joint disease is high in breast cancer patients. The cause of adhesive capsulitis is not clearly identified. However, the following are known as relevant factors that are the restriction of the use of the arm after surgery, inflammation due to autoimmune action, radiation therapy, and adhesion of the surgical site. The purpose of this study is to compare and analyze the effect of intrathecal steroid injection in breast cancer survivors with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent breast cancer surgery within 6 months.
* Patients with shoulder pain and limited range of motion

Exclusion Criteria:

* Patients with infection
* Bilateral shoulder pain patient
* Patients with uncontrolled diabetes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Range of motion of shoulder joint | Change from baseline at 3 months
  A goniometer is an instrument which measures the available range of motion at a joint.Flexion, Extension,Adduction,Abduction, Internal Rotation,External rotation

SECONDARY OUTCOMES:
Change in score on Shoulder Pain and Disability Index (SPADI) | Change from baseline at 3 months
  SPADI is a scale consisting of 0-10; 0 being the best and 10 being the worse pain ever; higher scores mean a worse outcome.
Axillary recess capsule thickness | Change from baseline at 3 months
  Ultrasound measurements of axillary recess capsule thickness in unilateral frozen shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Dong Gyu Dong Gyu, M.D., Ph.D., Principal Investigator — College of medicine, Yeungnam University
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No